CLINICAL TRIAL: NCT04995692
Title: Telehealth Education for Asthma Connecting Hospital and Home (TEACHH) Pilot Study
Brief Title: Telehealth Education for Asthma Connecting Hospital and Home
Acronym: TEACHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); American Lung Association (Other)
Responsible Party: Principal Investigator, Sean Frey, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00006450
Record Dates: First submitted 2021-07-14; First posted 2021-08-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Home Care Services; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial using a parallel design, in which subjects are randomized to one of two different arms
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting telephone follow-up assessments 2, 4, and 6 months after enrollment will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Education for Asthma Connecting Hospital and Home (TEACHH) (Experimental): New model of patient-centered asthma education
  Interventions: Behavioral: Telehealth Education for Asthma Connecting Hospital and Home
- Standard Care (SC) Comparison Group (Active Comparator): Standard inpatient asthma education per hospital protocol.
  Interventions: Behavioral: Standard Care (SC) Comparison Group

INTERVENTIONS:
Behavioral: Telehealth Education for Asthma Connecting Hospital and Home — TEACHH aims to provide educational support to families managing childhood asthma throughout the transition from hospital to home, and includes several core components: 1) Health literacy-informed inpatient teaching for child and caregiver including pictorial materials, hands-on demonstration, and use of teach-back/show-back techniques; 2) Facilitated identification of rescue and controller medications using color- and shape-coded medication labels and a pictorial asthma action plan; and 3) A pair of virtual follow-up visits after discharge to reinforce inpatient teaching and support families during the shift from acute exacerbation to preventive care management. Virtual visits will be completed using the Zoom platform on smartphones or other compatible devices, 2-4 days after discharge (first visit) and 3 weeks after discharge (second visit). All intervention activities will be completed within 1 month of discharge.
  Other Names: TEACHH
  Arms: Telehealth Education for Asthma Connecting Hospital and Home (TEACHH)
Behavioral: Standard Care (SC) Comparison Group — Patients in the SC group will receive standard impatient management, including pre-recorded asthma education videos shown prior to discharge and the hospital action plan. PCP follow-up with be scheduled within a week of discharge. All SC measures will also be provided to subjects randomized to TEACHH.
  Arms: Standard Care (SC) Comparison Group

SUMMARY:
The goal of this study is to evaluate the feasibility, acceptability, and preliminary efficacy of a technology-enhanced educational intervention for caregivers and children who are hospitalized due to asthma. We will conduct a pilot RCT with 60 children (5-13 yrs) hospitalized with asthma at the Golisano Children's Hospital in Rochester, NY. After baseline assessment, subjects will be randomized to either: 1) the Telehealth Education for Asthma Connecting Hospital and Home (TEACHH) intervention, which includes inpatient child/caregiver education using pictorial materials, color/shape labels for home medications (green star=controller, yellow/red circles=rescue), and a pair of in-home, smartphone-based telehealth visits after discharge to reinforce effective home management; or, 2) the standard care (SC) condition, which features standard inpatient education and routine outpatient follow-up. Patients in TEACHH will also receive all SC measures. All caregivers will complete blinded telephone follow-up assessments at 2, 4, and 6 months after discharge; children will be asked medication questions at baseline and 6 months. We will describe the feasibility and acceptability of implementing the TEACHH intervention by reviewing process measure data collected throughout the study; assess the preliminary efficacy of TEACHH in improving key clinical outcomes, including asthma-related ACU at 7 days, 30 days, and 6 months (per electronic health record documentation) and symptom-free days at each follow-up (reported by caregivers); and assess secondary clinical and functional outcomes including asthma-related quality of life, missed school or work due to asthma, caregiver and child medication knowledge, and reported adherence. We will also invite all caregivers to complete a semi-structured qualitative interview (1 month after baseline for the TEACHH group, 6 months after baseline for the SC group). Findings from this work will establish a strong foundation for a full-scale trial, and guide future efforts to deliver guideline-based asthma care to underserved children and families at the greatest risk for preventable morbidity.

DETAILED DESCRIPTION:
Study Design:

The investigators propose a 2-year pilot randomized trial of the TEACHH intervention vs. Standard Care (SC). We will enroll 60 children (5-13 years) with persistent asthma who are hospitalized at a tertiary care children's hospital with an acute asthma exacerbation. These children will be systematically screened, and those eligible approached for enrollment. After enrollment, participants will be randomly assigned to TEACHH or SC. We will measure feasibility continuously, and measure preliminary efficacy at 2, 4, and 6 months after enrollment. All caregivers will be invited to complete an additional in-depth interview to solicit feedback on the TEACHH intervention, and better understand family experiences with asthma management, educational support, and unmet home needs. We aim to conduct at least 20 interviews among caregivers in the TEACHH group, and 20 interviews among caregivers in the SC group.

Subjects and Setting:

Children aged 5-13 years will be screened for eligibility following admission to the Golisano Children's Hospital, a tertiary care institution in Rochester, NY. Eligibility will require persistent asthma severity (as per national guidelines) and a primary or secondary hospital diagnosis of asthma. We plan to enroll 60 children and caregiver dyads over a 12-month period. The mean length of stay at GCH for children with primary or secondary diagnoses of asthma is 3.8 days (1.9 days for primary diagnoses), ensuring ample time for study procedures. According to hospital census data, 386 children 5-13 years old with asthma are admitted for inpatient asthma care each year (128 primary diagnoses, 258 secondary diagnoses). We anticipate that at least 75% of these children (~290) will have persistent asthma symptoms and will be eligible for the pilot study, and we aim to enroll approximately 28% of the eligible children hospitalized within a 12-month timeframe.

These ages were chosen because: 1) younger children suffer the largest burden of asthma morbidity, 2) young children are at high risk for inadequate therapy for asthma, 3) children at age 5y are beginning to participate in medicine use, and 4) children in their mid-teenage have different medical and developmental needs compared to younger children, with different co-management roles with their parents that shift toward increased independence. The pictorial lessons, hands-on interactive demonstration of medication technique, and application of stickers to medications are all developmentally appropriate activities for this group of children.

Study Procedures:

Screening Procedures: Screening will occur in a rolling fashion from November 2021 through the end of October 2022. The investigators will identify potentially eligible children through a daily review of the inpatient census at the Golisano Children's Hospital. To be included in this study, children (5-13 years old) need to have (1) a physician diagnosis of asthma; (2) inpatient admission to the Golisano Children's Hospital with asthma as a primary or secondary diagnosis; and (3) persistent asthma or poor asthma control for which daily controller therapy is recommended by NHLBI guidelines. Caregivers will also need to have access to a smartphone (or similar device) for telehealth education. Dr. Frey will conduct a brief review of the patient's chart to determine whether key eligibility criteria are met (no known language barriers, no other significant medical or developmental conditions). Remaining eligibility criteria outlined above will be assessed during a brief screening visit with caregivers in the hospital.

Baseline Assessment: The baseline survey assessment will be conducted following enrollment by Dr. Frey or his research assistant within the child's hospital room or another comfortable, private inpatient setting. All survey instruments will be available in English, and questions will be read aloud to the caregiver and child. Although most questions will be posed to caregivers, children will also be asked several questions about their medications.

Randomization: After the baseline assessment, children will be randomly assigned to TEACHH or SC using a permuted block design to ensure an equal balance of children in each group over time. The URMC Biostatistics Center will develop the randomization scheme independently, and randomization will be implemented electronically via REDCapTM. All families will receive information on community resources for asthma management, addressing home asthma triggers, and smoking cessation. A letter describing study participation will be sent to each child's PCP.

TEACHH Intervention

Medicine Availability: All patients will have an albuterol MDI and spacer at the bedside per inpatient protocol. All subjects will have persistent asthma and should also be treated with a daily controller medication. We will ask inpatient providers to transmit controller prescriptions to the hospital outpatient pharmacy, which can send filled prescriptions to inpatient wards for labeling and teaching. If no prescriptions are needed, we will ask caregivers to bring controller medications from home. If controller medications are not available in the hospital, we will use practice inhalers for inpatient TEACHH activities and ensure proper medication labeling at the first virtual follow-up (below).

Inpatient asthma education, medication labeling, and smartphone set-up: A dedicated asthma educator will deliver inpatient education prior to discharge. We will use Zoom, an encrypted, HIPAA-compliant web-based program, for follow-up education and home management support. All major elements (teaching materials, medication labels, Zoom telehealth visits) have been successfully field tested. The inpatient session will include:

1. "Let's Take Control of Asthma," a brief, scripted overview of asthma, medications, and action plans that uses visual imagery to communicate essential teaching points.
2. Written information to support home management, including: a) pictorial instructions for using MDIs with a spacer; and b) a pictorial asthma action plan.
3. Color- and shape-coded stickers to distinguish controller and rescue medications (green star=controller, yellow/red circles=rescue). Labels will be applied by patients with caregiver assistance. Caregivers will apply matching labels to action plans for home reference when labeling refills. Additional labels will be provided for home. Teach-back will be used to ensure caregiver and child understanding of when to use each medicine.
4. A demonstration of correct technique for using inhaled medications. Teach-back and show-back methods will be used to verify comprehension.
5. Prior to discharge, the educator will help families download, install, and log in to Zoom from a smartphone or other available smart device (e.g., tablet).

Two videoconferencing sessions will be completed 2-4 days and 3 weeks after discharge by the same inpatient educator; timing will align with guideline recommendations for follow-up after hospitalization. Preferred times for visits will be reviewed prior to discharge. These visits are meant to supplement, not replace, recommended PCP follow-up visits.

First visit (2-4 days after discharge): This visit will reinforce key points of home management. The educator will show digital images from "Let's Take Control of Asthma," and review action plans, color/shape labels (including any medicines that were not available during hospitalization), and inhalation technique. Teach back will be used.

Second visit (3 weeks after discharge): This visit will emphasize ongoing management after an acute exacerbation, including continued use of controller medication and how to request and label refills. Session checklists will ensure that all components are delivered; ≥20% of sessions will be recorded and reviewed by the PI to assure fidelity and provide feedback.

Standard Care (SC) comparison condition:

Patients in the SC group will receive standard impatient management, including pre-recorded asthma education videos shown prior to discharge and the hospital action plan. PCP follow-up with be scheduled within a week of discharge. All SC measures will also be provided to subjects randomized to TEACHH.

Follow-Up Assessments:

The study, including all follow-up assessments, will continue throughout the 2022 calendar year and the first several months of 2023. We will follow subjects for a total of 6 months. After the baseline assessment, caregivers will complete 3 telephone-based surveys conducted 2-, 4-, and 6-months after discharge by a research assistant who is blinded to group allocation. Each assessment will repeat key measures from the baseline. We will use the electronic medical record (EMR) to review ACU and prescription fill data. To maintain blinding, we will not ask children about medications (indications for use, techniques) until the 6-month follow-up.

In-Depth Interviews:

Caregivers in both arms will also be invited to participate in semi-structured interviews. All caregivers will be eligible to participate in this, however we aim to complete 40 interviews altogether. The interview guide will explore family experiences with managing asthma at home, experiences with asthma education and management support before the index hospitalization, and caregiver opinions on support received during the index hospitalization with specific emphasis on components of the TEACHH intervention. Interviews will be conducted over Zoom (or by telephone if preferred), and audio recordings will be transcribed. Thematic analysis will be conducted on interview transcripts until saturation is achieved within both the TEACHH and SC groups; we anticipate completing 20 interviews in each group, that will take approximately 30-45 minutes to complete. In order to best capture feedback on the TEACHH intervention, we will interview caregivers randomized to this group approximately 1 month after enrollment (about 1 week after the second virtual visit). We plan to interview caregivers in the SC group after the final follow-up assessment, approximately 6 months after enrollment. During interviews with the SC group, we will show educational materials from the TEACHH intervention to solicit feedback.

ELIGIBILITY:
Inclusion Criteria (all 4 criteria must be met):

1. Physician diagnosis of asthma, based on review of medical records.
2. Inpatient admission to GCH with asthma as a primary or secondary diagnosis.
3. Persistent asthma or poor asthma control for which a daily controller medication is recommended by NHLBI guidelines, defined as any 1 of the following:

   1. >2 days per week with asthma symptoms in the past month;
   2. >2 days per week with rescue medication use in the past month;
   3. >2 days per month with nighttime symptoms in the past month; or
   4. ≥1 other episode(s) of asthma during the past year that required systemic corticosteroids
4. Age between ≥5 and ≤11 years.

Exclusion Criteria:

1. An inability to speak and understand English. Parents and children with low literacy / health-literacy skills will be eligible, as survey instruments will be administered verbally and educational materials will be designed for low-literacy populations.
2. No access to a working phone for follow-up survey assessments.
3. No access to a smartphone (or other 'smart' device) for telehealth education.
4. Another significant medical condition, including Cystic Fibrosis, congenital heart disease, or other chronic lung disease, that could interfere with assessment of asthma-related measures.
5. A diagnosed developmental condition (e.g. Autism spectrum disorder or significant developmental delay) identified in the child's medical record that could interfere with a child's ability to participate in teaching activities, and/or potentially delay the transition of responsibility for inhaled asthma medications from caregiver to child.
6. If the child or family is currently enrolled in a study conducted by The Preventive Care Program for Urban Children with Asthma (led by Dr. Jill Halterman).

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Asthma-related hospitalizations and emergency department visits after discharge | 7 days after discharge
  Asthma-related hospitalizations or emergency department visits, and drawn from objective healthcare utilization data in the electronic health record.
Asthma-related hospitalizations and emergency department visits after discharge | 30 days after discharge
  Asthma-related hospitalizations or emergency department visits, and drawn from objective healthcare utilization data in the electronic health record.
Asthma-related hospitalizations and emergency department visits after discharge | 6 months after discharge
  Asthma-related hospitalizations or emergency department visits, and drawn from objective healthcare utilization data in the electronic health record.
Symptom-Free Days (SFD) in the past 2 weeks | 2 months
  The number of 24-hour periods within the previous 14 days that a child remained free of asthma symptoms (range: 0-14 days); a higher score indicates more days without symptoms. Reported by caregivers during scheduled telephone assessments (2, 4, and 6 months after discharge)
Symptom-Free Days (SFD) in the past 2 weeks | 4 months
  The number of 24-hour periods within the previous 14 days that a child remained free of asthma symptoms (range: 0-14 days); a higher score indicates more days without symptoms. Reported by caregivers during scheduled telephone assessments (2, 4, and 6 months after discharge)
Symptom-Free Days (SFD) in the past 2 weeks | 6 months
  The number of 24-hour periods within the previous 14 days that a child remained free of asthma symptoms (range: 0-14 days); a higher score indicates more days without symptoms. Reported by caregivers during scheduled telephone assessments (2, 4, and 6 months after discharge)

SECONDARY OUTCOMES:
Caregiver-reported Asthma-related Acute Care Utilization (ACU) | 7 days, 30 days, and 6 months after discharge
  Asthma-related hospitalizations or emergency department visits; reported by caregivers during scheduled telephone assessments.
Caregiver-reported Asthma-related outpatient care | 2 months, 4 months, and 6 months
  Asthma-related visits to a primary care or urgent care clinic, including well-child checks in which asthma is managed; reported by caregivers during scheduled telephone assessments.
Caregiver-reported Asthma control (NHLBI) | 2 months, 4 months, and 6 months
  Asthma control over the past 1 month, as based on caregiver report of recent symptoms, activity limitation, and medication use during scheduled telephone assessments.
Caregiver quality of life | 2 months, 4 months, 6 months
  The Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) is a well-established, validated measure of caregiver quality of life over the previous 1 week, as reported by caregivers during scheduled telephone assessments (score range: 1-7 points; 1 indicates severe impairment, 7 indicates no impairment).
Missed school due to asthma in the past 2 weeks | 2 months, 4 months, 6 months
  We will ask caregivers to report how many days of school the child missed (if any) during the previous 2 weeks due to their asthma (range: 0-14 days).
Missed work due to asthma in the past 2 weeks | 2 months, 4 months, 6 months
  We will ask caregivers to report how many days of work the caregiver missed (if any) during the previous 2 weeks due to their child's asthma (range: 0-14 days).
Caregiver-reported Medication adherence | 2 months, 4 months, 6 months
  Recent adherence with prescribed controller therapy as reported by caregivers during scheduled telephone assessments using the Horne adherence scale (Score range: 40-20 points; higher scores indicate higher levels of reported adherence).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frey SM, Sanchez I, Fagnano M, Milne Wenderlich A, Mammen JR, Halterman JS. The Telehealth Education for Asthma Connecting Hospital and Home (TEACHH) pilot study. J Asthma. 2025 Mar;62(3):416-426. doi: 10.1080/02770903.2024.2408304. Epub 2024 Oct 9. PMID 39352693